CLINICAL TRIAL: NCT04679454
Title: Phase I/II Clinical Trial on Single Fraction Ablative Preoperative Radiation Treatment for Early Stage Breast Cancer
Brief Title: Single Fraction Preoperative Radiotherapy for Early Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 1308 - AIRC IG-23118
Record Dates: First submitted 2020-11-24; First posted 2020-12-22 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: preoperative radiotherapy; radiosurgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Radiation Treatment (Experimental): Preoperative Radiation treatment with CyberKnife
  Interventions: Radiation: Phase I; Radiation: Phase II

INTERVENTIONS:
Radiation: Phase I — To establish the recommended dose defined as the maximum tolerated dose (MTD)The dose-limiting toxicity (DLT) is defined as any G3-G4 event according to NCI CTCAE Version 4.03 scale. Dose escalation is designed as a 3+3 rule-based study. Dose escalation will be initiated from a baseline dose of 18 Gy and increased to reach 21 Gy and 24 Gy. The population size includes 18 patients.
Radiation: Phase II — The recommended dose from the phase I study is delivered, using Cyberknife in order to evaluate the efficacy measured in terms of pCR rate. The population size includes 61 patients.

SUMMARY:
This is a phase I/II, single-arm and open-label single-centre clinical trial with the aim to test the feasibility, safety and the efficacy, in terms of complete pathological response, of preoperative ablative radiotherapy in single fraction for selected breast cancer patients.

DETAILED DESCRIPTION:
The research plan is conceived in two sections, as follows. (i)The technical study handles the set-up, motion and dosimetric issues of the radioablation technique using CyberKnife system.

(ii)The clinical section is organized in two studies: a phase I dose escalation study to identify the maximum tolerated dose (MTD) delivering 18 Gy, 21 Gy and 24 Gy in single fraction and a phase II study to evaluate the rate of pathological complete response (pCR) when a dose level is chosen according to the results of the previous phase I study.

Study population includes patients affected by cT1-T2 (up to 2.5 cm) cN0, adenocarcinoma of the breast, diagnosed with conventional workup. Surgical tumor removal will be scheduled after 4-8 weeks after radioablation. Whole breast radiation therapy without boost will be performed after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven unifocal adenocarcinoma
* T1-T2
* Tumor size up to 2.5 cm
* cN0
* Age ≥ 18 years old
* Good general condition (ECOG 0-2)
* Planned BCS
* Written informed consent

Exclusion Criteria:

* Tumor close to skin or chest wall
* Pure non-invasive tumor
* Prior RT to the chest
* Neoadjuvant chemotherapy
* Collagenopathies
* Coagulation or autoimmunitary disorders
* Previous malignancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Phase I: Identify the maximum tolerated dose (MTD) | time frame:2 weeks
  Dose escalation is designed as a 3+3 rule-based study. Acute skin/soft tissue toxicity, measured according to NCI CTCAE v. 4.03. Any Grade 3-4 toxicity related to radioablation is considered dose limiting (DLT).
Phase II: Evaluate efficacy measured in terms of pCR rate | time frame:8 weeks
  Rate of pCR after radioablative treatment, according to Modified Residual Cancer Burden (RCB) index

SECONDARY OUTCOMES:
Incidence of chronic toxicity | time frame: 6 months - 3 years
  Chronic skin/soft tissue, bone, lung and heart toxicities incidence measured according to NCI CTCAE v. 4.03
Cosmetic outcomes | time frame: 1 - 3 years
  Measured according to the 4 points scale (poor, fair, good, excellent)
Post surgery complications | time frame: within 30 days of surgery
  Reporting of any post surgery complication (rate of infection, seroma, hematoma, necrosis, delayed wound healing)
Disease free survival | time frame: 1- 3 years
  establish the rate of disease free survival
Local relapse | time frame: 1 - 3 years
  establish the rate of local relapse
Overall survival | time frame: 3 years
  establish the rate of overall survival
Breast cancer specific survival | time frame: 3 years
  establish the rate of breast cancer specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Leonardi, Principal Investigator — European Institute of Oncology
Locations (1):
- IEO, European Institute of Oncology IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zerella MA, Zaffaroni M, Ronci G, Dicuonzo S, Rojas DP, Morra A, Gerardi MA, Fodor C, Rondi E, Vigorito S, Penco S, Sargenti M, Baratella P, Vicini E, Morigi C, Kahler-Ribeiro-Fontana S, Galimberti VE, Gandini S, De Camilli E, Renne G, Cattani F, Veronesi P, Orecchia R, Jereczek-Fossa BA, Leonardi MC. A narrative review for radiation oncologists to implement preoperative partial breast irradiation. Radiol Med. 2023 Dec;128(12):1553-1570. doi: 10.1007/s11547-023-01706-6. Epub 2023 Aug 31. PMID 37650981
- [Derived] Zerella MA, Zaffaroni M, Ronci G, Dicuonzo S, Rojas DP, Morra A, Fodor C, Rondi E, Vigorito S, Botta F, Cremonesi M, Garibaldi C, Penco S, Galimberti VE, Intra M, Gandini S, Barberis M, Renne G, Cattani F, Veronesi P, Orecchia R, Jereczek-Fossa BA, Leonardi MC. Single fraction ablative preoperative radiation treatment for early-stage breast cancer: the CRYSTAL study - a phase I/II clinical trial protocol. BMC Cancer. 2022 Apr 2;22(1):358. doi: 10.1186/s12885-022-09305-w. PMID 35366825